CLINICAL TRIAL: NCT05798988
Title: Neurophysiology-based Physiotherapy Program Effect on Selected Musculoskeletal Dysfunctions in Young Football Players
Brief Title: Physiotherapy Program Effect on Musculoskeletal Dysfunctions in Young Football Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jitka Marenčáková, Researcher, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UKFTVS_LSM_01
Record Dates: First submitted 2023-03-08; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Flatfoot, Flexible; Pes Valgus; Pes Varus; Balance; Distorted; Diastasis; Weak; Muscle
Keywords: Dynamic neuromuscular stabilisation; pronated foot; postural stability; neuromuscular control; exercise; sportive children; functional stabilisation; foot function; soccer
MeSH Terms: conditions — Flatfoot; Clubfoot; Asthenia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group will follow 8 weeks of neurophysiology-based exercise program.
  Interventions: Behavioral: Neurophysiology-based exercise program
- Control group (No Intervention): Control group will receive no intervention. They will not change the movement habits.

INTERVENTIONS:
Behavioral: Neurophysiology-based exercise program — Neurophysiology-based exercise program combines physiotherapy exercises and neuro-physiology principles with focus on foot and core functional stabilisation and balance training.
  Arms: Experimental group

SUMMARY:
The goal of this clinical study is to test the proposed physiotherapy exercise program in young football players. The main question it aims to answer is:

- Does the proposed physiotherapy program work well in improving young football players movement apparatus functions?

Participants will be asked to fill out questionaires about their musculoskeletal health, physical activity and foot wear and follow the 8 weeks of the group exercise program of 16 sessions in total (2 sessions per week, 30 minutes each session).

Researcher will compare exercising participants with no exercising participants of the same age and football category to see if the exercise program works well in young football players.

DETAILED DESCRIPTION:
The clinical trial aims to evaluate the short and long term effect of proposed neurophysiology-based physiotherapy program (NPP) on selected functional variables of the lower body in young football players, using clinical and laboratory diagnostic methods. Participants will be randomly assigned into one of the two groups: experimental (following 8 weeks of the intervention program) and control group (not changing the movement habits). Proposed NPP combines techniques and concepts based on neurophysiology principles and developmental kinesiology: sensorimotor stimulation and foot exercises, balance training, trunk stabilisation exercise in developmental kinesiology positions. Participants will exercise in small group twice a week in total of 16 sessions, 30 minutes each of session, under the guidance of an experienced physiotherapist. NPP is designed as a step by step progressive exercise program with focus on quality of neuromuscular control. Whole program is implemented into the standard football training process. Data will be obtained pre- (at baseline) and post-intervention (in 2 months and in 5 months) and compared to control group.

ELIGIBILITY:
Inclusion Criteria:

* participants playing football at sub- to elite level

Exclusion Criteria:

* acute infectious disease or fever
* any serious cardiological, neurological, or orthopedic diseases
* acute pain
* injury in the last 3 months
* currently undergoing any other kind of physiotherapy or treatment
* missing two or more sessions of the intervention program

Ages: 11 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Clinical foot type at 2 and 5 months | at baseline, in 2 months and in 5 months
  The foot posture will be assessed using the Foot posture index (6-FPI) evaluating six items (-2 and -1 for supination, 0 for neutral, and +1 and +2 for pronation) with final scores for 5 types of the foot: over-supinated foot (-12 to -5), supinated foot (-4 to -1), neutral foot (0 to +5), pronated foot (+6 to +9), and over-pronated foot (+10 to +12).
Change from baseline Calcaneal position in frontal plane at 2 and 5 months | at baseline, in 2 months and in 5 months
  The calcaneal position in frontal plane will be assessed using the Foot posture index (6-FPI) evaluating as one of the six items by points -2 and -1 for calcaneal inversion, 0 for neutral, and +1 and +2 for calcaneal eversion.
Change from baseline Medial longitudinal arch (MLA) height at 2 and 5 months | at baseline, in 2 months and in 5 months
  The MLA height will be assessed using the Foot posture index (6-FPI) evaluating as one of the six items by points -2 and -1 for calcaneal inversion, 0 for neutral, and +1 and +2 for calcaneal eversion.
Change from baseline Foot morphology at 2 and 5 months | at baseline, in 2 months and in 5 months
  The morphological parameters of the foot will be examined on a full foot 3D scanner (RSscan International, Belgium). A 3D image (scan) of the leg is obtained in two situations: sitting (10% weight-bearing) and resting (50% weight-bearing). In each situation, the proband remains still for the entire time of scanning (about 20 s).
  First, the measurement is performed while sitting, in a standardized position (90° flexion in the knee and ankle joint, shank vertical, sitting upright, hands on the hips). From a sitting position, the proband stands up in such a way that the weight of the body is distributed ideally evenly on both legs, upright calm standing, hands on the hips.
  From the obtained 3D data, parameters such as the foot length, foot width, and height of the MLA of the foot will be subtracted (mm).
Change from baseline Arch height index at 2 and 5 months | at baseline, in 2 months and in 5 months
  The Arch height index (AHI, %) will be calculated as the ratio of the dorsal MLA height measured at 50% of the truncated foot length and of the truncated foot length, in two positions: 1) AHI in sitting (10%WB) and 2) AHI in standing (50%WB).
Change from baseline Foot flexibility at 2 and 5 months | at baseline, in 2 months and in 5 months
  From the AHI values for sitting (10%WB) and for standing (50%WB) and body weight the Arch height flexibility (AHF, mm/kN) will be calculated. AHF evaluates the flexibility of the longitudinal arch independently on the clinical foot type. The basic results determine the flexibility of the foot as normal, rigid or flexible.
Change from baseline Postural stability at 2 and 5 months | at baseline, in 2 months and in 5 months
  The measurement will be provided using a pressure plate RS Footscan® (RSscan International, Paal, Belgium) with dimensions of 58x42x1.2 cm with a used imaging frequency of 10 Hz.
  The assessment will consist of narrow stance (NS) position and single-leg stance (SLS) position.
  1. The NS examination will be performed while standing in a narrow base first with eyes open and then with eyes closed for 33 seconds, with a pause of 30 seconds between the two conditions.
  2. The SLS testing will be performed while standing on the one leg for 60 seconds with repetition on the second leg. There will be a pause of 30 seconds between individual measurements.
  The parameter Centre of pressure path length (COPP) in millimeters and the maximum deviation achieved in the latero-lateral and antero-posterior directions in millimeters will be evaluated. The parameters are used to evaluate the level of postural stability of the individual.
Change from baseline Trunk stabilization function at 2 and 5 months | at baseline, in 2 months and in 5 months
  The trunk stabilization examination will be performed according to the examination protocol of the Dynamic Neuromuscular Stabilization (DNS) concept in the position from developmental ontogenesis - 3rd month lying on the back (Supine test). Evaluation of the quality of trunk stabilization: normal (0), impaired function (1), insufficient function with diastasis (2).

CONTACTS AND LOCATIONS:
Overall Officials: František Zahálka, prof., Ph.D., Study Director — Faculty of Physical Education and Sport, Charles University; Jitka Marenčáková, Ph.D., Principal Investigator — Faculty of Physical Eduction and Sport, Charles University
Locations (1):
- Faculty of Physical Education and Sport, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
It is planned that the anonymised data will be placed into an online repository (to be specified later)
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available after 6 months after the first publication for 2 years from the first publication.
Access Criteria: The datasets may be shared on the request and just on the basis of signed Data-Sharing Agreement between the new user and research team. The study team formally reviews access requests for proposals. The use of the datasets by third party can range from direct provision of data, to data analysis collaboration, and/or scientific collaboration.